CLINICAL TRIAL: NCT00125463
Title: Candesartan Antihypertensive Survival Evaluation in Japan (CASE-J) Trial of Cardiovascular Events in High-Risk Hypertensive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Japanese Society of Hypertension (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSH-00001
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2005-08-10 (Estimated); Status verified 2005-04

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Hypertension; clinical trial; Candesartan Antihypertensive Survival Evaluation in Japan trial; candesartan cilexetil; amlodipine besilate
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — candesartan cilexetil

INTERVENTIONS:
Drug: Candesartan cilexetil

SUMMARY:
The purpose of this study is to compare an angiotensin II receptor antagonist (candesartan cilexetil- Blopress®) and a calcium channel blocker (amlodipine besilate- Norvasc®/Amlodin®) in terms of the incidence of cardiovascular events among high-risk hypertensive patients.

DETAILED DESCRIPTION:
Hypertension continues to be a major public health issue in the world. To combat this problem, many antihypertensive drugs have been developed and proven effective at controlling blood pressure in the last half century. In recent decades, antihypertensive drugs have been shown to have cardiovascular benefits beyond the reduction of blood pressure, and the focus has shifted to clarification of these effects. Angiotensin II receptor antagonists and calcium channel blockers are the most widely used antihypertensive drugs in Japan. However, these two classes of drugs have not yet been compared with respect to their efficacy for treating cardiovascular events.

Comparison: Response-dependent dose titration and blinded assessment of endpoints in high risk hypertensive patients treated with either an angiotensin II receptor antagonist (candesartan cilexetil) compared to a third-generation calcium channel blocker (amlodipine besilate).

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP) ≥140 mmHg in those <70 years old or ≥160 mmHg in those ≥70 years old or diastolic blood pressure (DBP) ≥90 mmHg in a sitting position on two consecutive measurements at clinic
* At least one of the following risk factors:

  * SBP ≥180 mmHg or DBP ≥110 mmHg on two consecutive visits;
  * Type 2 diabetes (fasting blood glucose ≥126 mg/dl, causal blood glucose ≥200 mg/dl, HbA1c ≥6.5%, 2 hours blood glucose on 75 g oral glucose tolerance test [OGTT] ≥200 mg/dl, or current treatment with hypoglycemic agent);
  * History of cerebral hemorrhage, cerebral infarction, or transient ischemic attack until 6 months prior to the screening;
  * Thickness of the posterior wall of left ventricle or thickness of the wall of interventricular septum ≥12 mm on echocardiography or Sv1＋Rv5 ≥35 mm on electrocardiography, angina pectoris, and a past history (≥6 months before giving informed consent) of myocardial infarction;
  * Proteinuria ≥＋1 or renal impairment (serum creatinine ≥1.3 mg/dl) within 3 months at the time of giving informed consent;
  * Arteriosclerotic peripheral arterial obstruction (Fontaine class ≥2); *Clinical diagnosis of Alzheimer's disease.

Exclusion Criteria:

* SBP ≥200 mmHg or DBP ≥120 mmHg in a sitting position
* Type I diabetes mellitus
* History of myocardial infarction or cerebrovascular accidents within 6 months prior to the screening
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass grafting (CABG) done within 6 months of screening or scheduled
* Current treatment for congestive cardiac failure (New York Heart Association [NYHA] functional class II or severer) or ejection fraction <40%
* Coronary artery disease requiring αβ blocker or calcium channel blocker
* Atrial fibrillation or atrial flutter
* Renal dysfunction (serum creatinine ≥3 mg/dl)
* Hepatic dysfunction (AST and/or ALT ≥100 IU/l)
* A history of malignant tumor within 5 years of enrollment or suspected
* Contraindication for candesartan cilexetil or amlodipine besilate
* Pregnancy, possible pregnancy, or plan to conceive a child within 5 years of enrollment
* Not suited to the clinical trial as judged by a collaborating physician
* Inability to give informed consent

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Start 2001-09; Study Completion 2005-12

PRIMARY OUTCOMES:
Sudden death: death of endogenous origin within 24 hours after acute onset
Cerebrovascular events: new occurrence or recurrence of a stroke or transient ischemic attack
Cardiac events: new occurrence, aggravation, or recurrence of heart failure, angina pectoris, or acute myocardial infarction
Renal dysfunction: serum creatinine ≥4.0 mg/dl, end stage renal disease, doubling of serum creatinine (however, creatinine ≤2.0 mg/dl is not regarded as an event)
Vascular events: new occurrence or aggravation of dissecting aneurysm of aorta, arteriosclerotic occlusion of peripheral artery

SECONDARY OUTCOMES:
All deaths
Involution of left ventricular hypertrophy (LVMI)
Proportion of the subjects who withdrew from the allocated treatment

CONTACTS AND LOCATIONS:
Overall Officials: Takao Saruta, M.D., Principal Investigator — Keio University
Locations (1):
- Kyoto University, Kyoto, Yoshidakonoe-cho, Sakyo-ku, Kyoto, Japan

REFERENCES:
- [Background] Fukui T, Rahman M, Hayashi K, Takeda K, Higaki J, Sato T, Fukushima M, Sakamoto J, Morita S, Ogihara T, Fukiyama K, Fujishima M, Saruta T; CASE-J Study Group. Candesartan Antihypertensive Survival Evaluation in Japan (CASE-J) trial of cardiovascular events in high-risk hypertensive patients: rationale, design, and methods. Hypertens Res. 2003 Dec;26(12):979-90. doi: 10.1291/hypres.26.979. PMID 14717341
- [Derived] Ogihara T, Nakao K, Fukui T, Fukiyama K, Fujimoto A, Ueshima K, Oba K, Shimamoto K, Matsuoka H, Saruta T; CASE-J Trial Group. The optimal target blood pressure for antihypertensive treatment in Japanese elderly patients with high-risk hypertension: a subanalysis of the Candesartan Antihypertensive Survival Evaluation in Japan (CASE-J) trial. Hypertens Res. 2008 Aug;31(8):1595-601. doi: 10.1291/hypres.31.1595. PMID 18971535